CLINICAL TRIAL: NCT01923480
Title: Determination of the Optimal Infusion Rate of Amino Acids in Seriously Ill Patients
Brief Title: Dosing Study of Amino Acids in Seriously Ill Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CT-12-0012
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Results first posted 2017-03-27 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2016-02

CONDITIONS: Parenteral Nutrition (No Primary Condition Studied)
MeSH Terms: conditions — Hyperphagia | interventions — Amino Acids; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 15% CLINISOL 0.04 g/kg/hr (Experimental): 15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.04 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection.
  Interventions: Drug: 15% CLINISOL - Sulfite-free (Amino Acid) Injection
- 15% CLINISOL 0.08 g/kg/hr (Experimental): 15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.08 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection.
  Interventions: Drug: 15% CLINISOL - Sulfite-free (Amino Acid) Injection
- 15% CLINISOL 0.13 g/kg/hr (Experimental): 15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.13 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection.
  Interventions: Drug: 15% CLINISOL - Sulfite-free (Amino Acid) Injection

INTERVENTIONS:
Drug: 15% CLINISOL - Sulfite-free (Amino Acid) Injection
  Arms: 15% CLINISOL 0.04 g/kg/hr
Drug: 15% CLINISOL - Sulfite-free (Amino Acid) Injection
  Arms: 15% CLINISOL 0.08 g/kg/hr
Drug: 15% CLINISOL - Sulfite-free (Amino Acid) Injection
  Arms: 15% CLINISOL 0.13 g/kg/hr

SUMMARY:
The purpose of this study is to determine the best rate of infusion of amino acids (15% CLINISOL - sulfite-free (Amino Acid) Injection) for nutrition in subjects with with stages II to IVB head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Have Stages II to IVB head and neck cancer receiving radiation and may also be receiving chemotherapy.

  * Subjects are eligible for inclusion in the study regardless of primary Stages II to IVB head and neck cancer treatment modality (eg, surgery, chemotherapy).
* Have voluntarily signed and dated a written informed consent form (ICF) after the nature of the study was explained to them.
* Female subjects must be of non childbearing potential (defined as postmenopausal for at least 1 year or surgically sterile [bilateral tubal ligation, bilateral oophorectomy or hysterectomy]) or;
* Female subjects of childbearing potential must be using adequate contraception (practicing 1 of the following methods of birth control):

  * total abstinence from sexual intercourse (minimum of 1 complete menstrual cycle before study entry),
  * a vasectomized partner,
  * contraceptives (oral, parenteral, or transdermal) for 3 consecutive months prior to study drug administration,
  * intrauterine device (IUD), or
  * double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream).
* Female subjects must have a negative serum or urinary pregnancy test result at screening (serum specimen must be obtained within 14 days prior to baseline).

Exclusion Criteria:

* Had a loss of > 10% of body weight within the 3 month period prior to the study as noted in the subjects medical history chart.
* Have renal disease as determined by an estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2.
* Have a hemoglobin level of < 9 g/dl.
* Have Stage 0, I, or IVC metastatic cancer.
* Have diabetes.
* Have any reason which, in the opinion of the Investigator, would prevent the subject from safely participating in the study.
* Have, in the opinion of the Investigator, a dependence on alcohol.
* Have, in the opinion of the Investigator, a dependence on illicit drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Texas A&M University, Center for Translational Research in Aging & Longevity, College Station, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- 15% CLINISOL 0.04 g/kg/hr (AB): Sequence AB - without Insulin first, then with insulin
  15% CLINISOL- Sulfite-Free (Amino Acid) Injection 0.04 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection
- 15% CLINISOL 0.04 g/kg/hr (BA): Sequence BA - with Insulin first, then no insulin
  15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.04 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection
- 15% CLINISOL 0.08 g/kg/hr (AB): Sequence AB - without Insulin first, then with insulin
  15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.08 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection
- 15% CLINISOL 0.08 g/kg/hr (BA): Sequence BA - with Insulin first, then no insulin
  15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.08 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection
- 15% CLINISOL 0.13 g/kg/hr (AB): Sequence AB - without Insulin first, then with insulin
  15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.13 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection
- 15% CLINISOL 0.13 g/kg/hr (BA): Sequence BA - with Insulin first, then no insulin
  15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.13 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection
Period: Period 1 (Hours 1-7)
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Started | 1 | 2 | 2 | 2 | 2 | 2
Completed | 1 | 2 (One subject completed Period 1, but withdrew from the study prior to the start of Period 2.) | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Hours 1-7)
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Started | 1 | 1 (One subject completed Period 1, but withdrew from the study prior to the start of Period 2.) | 2 | 2 | 2 | 2
Completed | 1 | 1 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 15% CLINISOL 0.04 g/kg/hr: 15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.04 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection.
  15% CLINISOL - Sulfite-free (Amino Acid) Injection
- 15% CLINISOL 0.08 g/kg/hr: 15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.08 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection.
  15% CLINISOL - Sulfite-free (Amino Acid) Injection
- 15% CLINISOL 0.13 g/kg/hr: 15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.13 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection.
  15% CLINISOL - Sulfite-free (Amino Acid) Injection
- Total: Total of all reporting groups
Arm/Group | 15% CLINISOL 0.04 g/kg/hr | 15% CLINISOL 0.08 g/kg/hr | 15% CLINISOL 0.13 g/kg/hr | Total
Number analyzed (Participants) | 3 | 4 | 4 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at informed consent.
  Years | 60.33 (10.50) | 69.25 (14.93) | 60.50 (6.40) | 63.64 (11.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 1 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Net Protein Synthesis
Time Frame: One time at pre-clinisol infusion and one time at post-clinisol infusion
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: g protein/d/kg ffm
Groups:
- 15% CLINISOL 0.04 g/kg/hr (AB): Sequence AB - without Insulin first, then with Insulin
  15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.04 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid) Injection
- 15% CLINISOL 0.08 g/kg/hr (BA): Sequence BA - with Insulin first, then no Insulin
  15% CLINISOL- Sulfite-Free (Amino Acid)Injection 0.08 g/kg/hr to be administered. Each treatment session is expected to last 7 hours with the first 3 hours of basal infusion followed by 4 hours of 15% CLINISOL - Sulfite-Free (Amino Acid)
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
g protein/d/kg ffm
  Period 1 | 2.82 (0) | 3.15 (0.38) | 4.92 (0.45) | 11.62 (6.67) | 6.11 (2.46) | 9.15 (2.64)
  Period 2: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 | 2.6 (0) | 2.83 (0) | 6.13 (0.62) | 4.89 (0.81) | 9.10 (2.52) | 8.29 (0.88)

2. Secondary Outcome: Insulin Sensitivity
Time Frame: Five times during each 7 hour visit
Population: No data available as no data for this outcome measure were collected during the study.
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Plasma Concentration of Glucose
Time Frame: Nine times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2. One subject in grp 0.04 g/kg/hr, seq BA, plasma concentration of glucose was not collected at any time point during Period 1.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
mg/dL
  Period 1 @ 3hrs | 101.0 (0) | 92.00 (0) | 90.00 (4.24) | 93.50 (2.12) | 102.0 (21.21) | 95.00 (7.07)
  Period 1 @ 3.5hrs | 101.0 (0) | 81.00 (0) | 93.00 (5.66) | 94.00 (8.49) | 104.0 (19.80) | 111.5 (7.78)
  Period 1 @ 4hrs | 100.0 (0) | 91.00 (0) | 94.00 (5.66) | 97.00 (1.41) | 103.5 (13.44) | 110.0 (15.56)
  Period 1 @ 4.5hrs | 93.00 (0) | 102.0 (0) | 96.50 (3.54) | 90.00 (12.73) | 107.50 (14.85) | 105.5 (7.78)
  Period 1 @ 5hrs | 95.00 (0) | 111.0 (0) | 94.50 (3.54) | 92.50 (7.78) | 104.5 (13.44) | 95.50 (9.19)
  Period 1 @ 5.5hrs | 93.00 (0) | 89.00 (0) | 95.00 (1.41) | 97.00 (11.31) | 101.0 (15.56) | 96.50 (9.19)
  Period 1 @ 6hrs | 97.00 (0) | 75.00 (0) | 93.00 (1.41) | 98.00 (1.41) | 105.5 (14.85) | 93.50 (9.19)
  Period 1 @ 6.5hrs | 99.00 (0) | 69.00 (0) | 93.00 (1.41) | 92.50 (3.54) | 100.0 (11.31) | 95.00 (7.78)
  Period 1 @ 7hrs | 97.00 (0) | 99.00 (0) | 91.50 (2.12) | 86.50 (0.71) | 101.5 (14.85) | 93.50 (2.12)
  Period 2 @ 3hrs | 95.00 (0) | 102.0 (0) | 88.00 (2.83) | 96.00 (4.24) | 102.5 (20.51) | 94.50 (9.19)
  Period 2 @ 3.5hrs | 103.00 (0) | 97.00 (0) | 88.00 (32.53) | 101.0 (5.66) | 99.00 (45.25) | 100.0 (8.49)
  Period 2 @ 4hrs | 103.0 (0) | 104.0 (0) | 90.50 (28.99) | 99.50 (4.95) | 100.5 (37.48) | 103.5 (6.36)
  Period 2 @ 4.5hrs | 108.0 (0) | 103.0 (0) | 92.00 (9.90) | 98.00 (1.41) | 103.0 (26.87) | 100.0 (7.07)
  Period 2 @ 5hrs | 110.0 (0) | 103.00 (0) | 95.00 (8.49) | 99.00 (4.24) | 104.5 (19.09) | 100.0 (9.90)
  Period 2 @ 5.5hrs | 103.00 (0) | 104.0 (0) | 90.50 (6.36) | 98.00 (1.41) | 112.5 (7.78) | 101.5 (10.61)
  Period 2 @ 6hrs | 97.00 (0) | 106.0 (0) | 93.00 (9.90) | 105.0 (7.07) | 105.0 (4.24) | 100.0 (8.49)
  Period 2 @ 6.5hrs | 86.00 (0) | 102.0 (0) | 84.50 (4.95) | 103.5 (6.36) | 101.5 (9.19) | 98.00 (8.49)
  Period 2 @ 7hrs | 86.00 (0) | 105.0 (0) | 75.00 (2.83) | 100.5 (0.71) | 107.0 (1.41) | 98.50 (10.61)

4. Secondary Outcome: Serum Concentration of Insulin
Time Frame: Five times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2. One subject in grp 0.04 g/kg/hr, seq BA, serum concentration of insulin was not collected at any time point during Period 1. One subject in grp 0.08 g/kg/hr, seq AB, serum concentration of insulin was not collected at the 3hr time point during Period 2.
Measure: Mean (Standard Deviation); unit: mciu/mL
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
mciu/mL
  Period 1 @ 3hrs | 13.70 (0) | 4.70 (0) | 14.10 (13.29) | 9.95 (1.20) | 6.90 (5.80) | 27.10 (19.37)
  Period 1 @ 4hrs | 23.50 (0) | 60.90 (0) | 19.10 (20.36) | 105.2 (0.78) | 12.60 (7.50) | 301.9 (206.9)
  Period 1 @ 5hrs | 21.80 (0) | 63.40 (0) | 21.65 (23.41) | 102.0 (7.50) | 12.10 (4.95) | 259.6 (194.3)
  Period 1 @ 6hrs | 24.40 (0) | 70.70 (0) | 20.95 (20.01) | 100.9 (11.17) | 9.05 (5.30) | 239.4 (192.3)
  Period 1 @ 7hrs | 20.80 (0) | 64.90 (0) | 16.60 (17.68) | 92.75 (26.09) | 9.35 (6.58) | 188.5 (128.9)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 1 | 2 | 2 | 2
  Period 2 @ 3hrs | 7.60 (0) | 7.80 (0) | 2.10 (0) | 7.40 (0.28) | 8.25 (2.05) | 66.20 (75.24)
  Period 2 @ 4hrs | 87.20 (0) | 7.20 (0) | 66.50 (4.95) | 15.30 (0.71) | 75.95 (23.55) | 139.3 (154.1)
  Period 2 @ 5hrs | 102.4 (0) | 5.10 (0) | 60.95 (1.63) | 12.15 (1.77) | 69.85 (9.26) | 168.8 (206.0)
  Period 2 @ 6hrs | 73.20 (0) | 5.80 (0) | 67.20 (8.49) | 17.65 (9.26) | 73.55 (6.15) | 173.0 (221.7)
  Period 2 @ 7hrs | 90.20 (0) | 7.90 (0) | 67.90 (12.16) | 13.15 (4.03) | 74.30 (15.41) | 143.0 (185.5)

5. Secondary Outcome: Plasma Stable Isotope Enrichment of Phenylalanine
Time Frame: Twelve times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2. During both periods (1 and 2), samples were not obtained from any subjects at the 0hr time point.
Measure: Mean (Standard Deviation); unit: trace/tracee ratio
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
trace/tracee ratio
  Period 1 @ 0hrs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Period 1 @ 2hrs | 0.14 (0) | 0.11 (0.01) | 0.09 (0.05) | 0.08 (0.09) | 0.10 (0.01) | 0.12 (0.01)
  Period 1 @ 2.5hrs | 0.15 (0) | 0.11 (0.01) | 0.09 (0.05) | 0.08 (0.10) | 0.12 (0.01) | 0.12 (0.01)
  Period 1 @ 3hrs | 0.16 (0) | 0.12 (0.01) | 0.10 (0.05) | 0.08 (0.10) | 0.11 (0.01) | 0.12 (0.02)
  Period 1 @ 3.5hrs | 0.13 (0) | 0.12 (0.01) | 0.09 (0.05) | 0.10 (0.05) | 0.11 (0.04) | 0.49 (0.56)
  Period 1 @ 4hrs | 0.12 (0) | 0.11 (0.01) | 0.09 (0.03) | 0.12 (0.04) | 0.12 (0.04) | 0.09 (0)
  Period 1 @ 4.5hrs | 0.12 (0) | 0.12 (0.01) | 0.10 (0.03) | 0.12 (0.04) | 0.12 (0.03) | 0.09 (0)
  Period 1 @ 5hrs | 0.12 (0) | 0.12 (0.01) | 0.10 (0.03) | 0.12 (0.04) | 0.12 (0.03) | 0.09 (0)
  Period 1 @ 5.5hrs | 0.12 (0) | 0.12 (0.01) | 0.09 (0.02) | 0.12 (0.04) | 0.12 (0.03) | 0.09 (0.01)
  Period 1 @ 6hrs | 0.11 (0) | 0.12 (0.01) | 0.10 (0.03) | 0.12 (0.04) | 0.12 (0.03) | 0.10 (0)
  Period 1 @ 6.5hrs | 0.12 (0) | 0.12 (0.01) | 0.10 (0.03) | 0.12 (0.04) | 0.14 (0.01) | 0.10 (0)
  Period 1 @ 7hrs | 0.12 (0) | 0.12 (0.01) | 0.08 (0.01) | 0.13 (0.04) | 0.13 (0.03) | 0.10 (0.01)
  Period 2 @ 0hrs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Period 2 @ 2hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 2hrs | 0.16 (0) | 0.09 (0) | 0.10 (0.04) | 0.13 (0) | 0.09 (0) | 0.10 (0.01)
  Period 2 @ 2.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 2.5hrs | 0.16 (0) | 0.10 (0) | 0.11 (0.04) | 0.14 (0.01) | 0.11 (0.01) | 0.11 (0.01)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 0.17 (0) | 0.10 (0) | 0.11 (0.04) | 0.14 (0.03) | 0.13 (0.01) | 0.12 (0.01)
  Period 2 @ 3.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3.5hrs | 0.14 (0) | 0.11 (0) | 0.10 (0.04) | 0.13 (0.02) | 0.10 (0.01) | 0.09 (0.01)
  Period 2 @ 4hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4hrs | 0.13 (0) | 0.11 (0) | 0.10 (0.03) | 0.12 (0.02) | 0.09 (0.01) | 0.09 (0)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 0.14 (0) | 0.12 (0) | 0.09 (0.03) | 0.12 (0.02) | 0.10 (0.01) | 0.09 (0)
  Period 2 @ 5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 5hrs | 0.15 (0) | 0.11 (0) | 0.10 (0.03) | 0.12 (0.02) | 0.10 (0.01) | 0.09 (0)
  Period 2 @ 5.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 5.5hrs | 0.14 (0) | 0.12 (0) | 0.10 (0.03) | 0.12 (0.02) | 0.10 (0.01) | 0.09 (0.01)
  Period 2 @ 6hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 6hrs | 0.15 (0) | 0.11 (0) | 0.10 (0.03) | 0.12 (0.02) | 0.10 (0.01) | 0.09 (0.01)
  Period 2 @ 6.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 6.5hrs | 0.15 (0) | 0.11 (0) | 0.10 (0.03) | 0.12 (0.02) | 0.10 (0.01) | 0.09 (0.01)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 0.16 (0) | 0.11 (0) | 0.10 (0.03) | 0.12 (0.02) | 0.10 (0.01) | 0.09 (0)

6. Secondary Outcome: Plasma Stable Isotope Enrichment of Tyrosine
Time Frame: Twelve times during each 7 hour visit
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: trace/tracee ratio
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
trace/tracee ratio
  Period 1 @ 0hrs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Period 1 @ 2hrs | 0.06 (0) | 0.03 (0.02) | 0.05 (0.02) | 0.07 (0.01) | 0.05 (0) | 0.08 (0.03)
  Period 1 @ 2.5hrs | 0.06 (0) | 0.03 (0.02) | 0.05 (0.02) | 0.07 (0.01) | 0.06 (0) | 0.08 (0.03)
  Period 1 @ 3hrs | 0.07 (0) | 0.04 (0.02) | 0.05 (0.02) | 0.07 (0.01) | 0.06 (0) | 0.09 (0.03)
  Period 1 @ 3.5hrs | 0.07 (0) | 0.04 (0.02) | 0.05 (0.02) | 0.08 (0.02) | 0.06 (0) | 0.08 (0.03)
  Period 1 @ 4hrs | 0.07 (0) | 0.04 (0.02) | 0.05 (0.02) | 0.08 (0.03) | 0.06 (0) | 0.08 (0.04)
  Period 1 @ 4.5hrs | 0.07 (0) | 0.04 (0.02) | 0.06 (0.02) | 0.08 (0.03) | 0.06 (0) | 0.09 (0.04)
  Period 1 @ 5hrs | 0.08 (0) | 0.05 (0.02) | 0.06 (0.02) | 0.09 (0.04) | 0.06 (0) | 0.09 (0.03)
  Period 1 @ 5.5hrs | 0.08 (0) | 0.04 (0.02) | 0.06 (0.02) | 0.09 (0.03) | 0.06 (0) | 0.09 (0.04)
  Period 1 @ 6hrs | 0.07 (0) | 0.05 (0.02) | 0.06 (0.02) | 0.09 (0.04) | 0.06 (0) | 0.09 (0.04)
  Period 1 @ 6.5hrs | 0.08 (0) | 0.05 (0.02) | 0.06 (0.02) | 0.10 (0.05) | 0.06 (0.01) | 0.09 (0.04)
  Period 1 @ 7hrs | 0.08 (0) | 0.05 (0.02) | 0.06 (0.02) | 0.10 (0.05) | 0.06 (0.01) | 0.09 (0.04)
  Period 2 @ 0hrs: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Period 2 @ 2hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 2hrs | 0.08 (0) | 0.04 (0) | 0.05 (0.02) | 0.06 (0.02) | 0.04 (0.01) | 0.07 (0.03)
  Period 2 @ 2.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 2.5hrs | 0.08 (0) | 0.05 (0) | 0.05 (0.01) | 0.07 (0.02) | 0.05 (0) | 0.08 (0.04)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 0.09 (0) | 0.05 (0) | 0.05 (0.01) | 0.07 (0.03) | 0.06 (0.01) | 0.08 (0.04)
  Period 2 @ 3.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3.5hrs | 0.08 (0) | 0.05 (0) | 0.06 (0.02) | 0.08 (0.03) | 0.05 (0.01) | 0.07 (0.03)
  Period 2 @ 4hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4hrs | 0.08 (0) | 0.05 (0) | 0.06 (0.01) | 0.08 (0.03) | 0.05 (0.01) | 0.08 (0.04)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 0.88 (0) | 0.05 (0) | 0.05 (0.01) | 0.08 (0.03) | 0.06 (0.01) | 0.08 (0.04)
  Period 2 @ 5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 5hrs | 0.09 (0) | 0.05 (0) | 0.06 (0.02) | 0.08 (0.03) | 0.06 (0.01) | 0.08 (0.04)
  Period 2 @ 5.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 5.5hrs | 0.09 (0) | 0.05 (0) | 0.06 (0.02) | 0.08 (0.03) | 0.06 (0.01) | 0.09 (0.05)
  Period 2 @ 6hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 6hrs | 0.09 (0) | 0.05 (0) | 0.06 (0.01) | 0.08 (0.04) | 0.06 (0.01) | 0.08 (0.04)
  Period 2 @ 6.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 6.5hrs | 0.09 (0) | 0.05 (0) | 0.06 (0.02) | 0.08 (0.04) | 0.06 (0.01) | 0.08 (0.04)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 0.10 (0) | 0.05 (0) | 0.06 (0.02) | 0.08 (0.04) | 0.06 (0.01) | 0.08 (0.04)

7. Secondary Outcome: Plasma Concentration of Alanine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 364.9 (0) | 239.6 (2.09) | 212.4 (7.83) | 321.5 (3.85) | 284.8 (199.2) | 428.2 (63.00)
  Period 1 @ 4.5hrs | 499.1 (0) | 292.9 (36.73) | 347.5 (3.14) | 648.9 (73.64) | 468.1 (195.4) | 840.3 (304.2)
  Period 1 @ 7hrs | 440.0 (0) | 359.6 (46.67) | 388.9 (10.32) | 645.1 (126.4) | 414.4 (101.8) | 959.3 (481.3)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 340.6 (0) | 425.8 (0) | 240.5 (8.59) | 449.5 (221.3) | 346.1 (266.3) | 522.7 (258.7)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 438.3 (0) | 407.1 (0) | 414.4 (86.71) | 813.7 (269.6) | 631.5 (292.7) | 938.9 (436.0)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 452.0 (0) | 463.3 (0) | 425.8 (11.01) | 770.3 (254.9) | 573.0 (209.0) | 976.6 (483.5)

8. Secondary Outcome: Plasma Concentration of Arginine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 98.48 (0) | 69.25 (11.33) | 71.35 (17.40) | 61.34 (2.09) | 82.74 (39.22) | 88.24 (5.66)
  Period 1 @ 4.5hrs | 153.8 (0) | 88.42 (22.85) | 145.8 (28.74) | 160.1 (13.87) | 171.9 (16.72) | 276.6 (75.96)
  Period 1 @ 7hrs | 160.5 (0) | 94.35 (3.58) | 159.7 (27.81) | 173.2 (2.28) | 167.8 (6.87) | 307.9 (108.7)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 84.17 (0) | 81.10 (0) | 85.71 (30.99) | 72.54 (7.09) | 79.34 (29.04) | 100.7 (22.21)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 120.4 (0) | 115.7 (0) | 151.6 (34.59) | 195.6 (9.68) | 204.1 (99.12) | 284.2 (86.42)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 130.3 (0) | 139.0 (0) | 152.7 (9.45) | 221.9 (36.78) | 200.9 (102.1) | 294.3 (86.06)

9. Secondary Outcome: Plasma Concentration of Aspartic Acid
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 3.98 (0) | 1.95 (0.39) | 2.18 (0.61) | 2.53 (0.12) | 2.88 (0.17) | 3.27 (0.66)
  Period 1 @ 4.5hrs | 10.47 (0) | 4.13 (2.79) | 9.52 (2.68) | 9.60 (0.67) | 12.56 (1.12) | 23.45 (1.58)
  Period 1 @ 7hrs | 10.95 (0) | 2.43 (0.59) | 9.24 (0.57) | 9.04 (3.01) | 9.73 (0.98) | 31.28 (11.53)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 2.87 (0) | 2.52 (0) | 2.40 (1.03) | 2.92 (0.55) | 3.71 (1.35) | 3.76 (1.28)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 7.57 (0) | 4.21 (0) | 6.55 (1.89) | 11.67 (0.36) | 15.38 (4.19) | 22.67 (0.95)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 7.99 (0) | 4.07 (0) | 8.98 (8.13) | 11.11 (1.20) | 15.43 (2.30) | 21.79 (0.23)

10. Secondary Outcome: Plasma Concentration of Glutamic Acid
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 586.0 (0) | 659.1 (120.1) | 561.1 (108.5) | 678.3 (28.45) | 588.4 (172.6) | 644.8 (27.42)
  Period 1 @ 4.5hrs | 634.8 (0) | 599.5 (167.4) | 561.9 (179.0) | 647.9 (48.97) | 646.6 (158.3) | 690.9 (100.7)
  Period 1 @ 7hrs | 647.8 (0) | 661.2 (93.35) | 573.7 (131.0) | 560.1 (99.21) | 576.0 (98.2) | 710.8 (211.5)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 587.3 (0) | 884.3 (0) | 588.9 (138.8) | 722.5 (125.8) | 607.5 (119.3) | 727.1 (153.3)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 510.8 (0) | 926.7 (0) | 563.5 (150.4) | 811.7 (159.9) | 606.9 (111.6) | 809.3 (180.6)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 489.2 (0) | 854.5 (0) | 510.0 (123.1) | 735.0 (215.9) | 531.4 (72.39) | 808.6 (237.8)

11. Secondary Outcome: Plasma Concentration of Glutamine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 75.20 (0) | 25.55 (11.72) | 43.94 (15.40) | 46.75 (0.04) | 60.22 (29.73) | 69.89 (18.67)
  Period 1 @ 4.5hrs | 99.73 (0) | 25.08 (1.92) | 70.98 (27.55) | 65.68 (2.20) | 105.1 (38.45) | 142.3 (18.79)
  Period 1 @ 7hrs | 100.0 (0) | 18.58 (5.77) | 68.48 (14.21) | 60.20 (17.41) | 92.00 (25.10) | 175.10 (30.72)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 71.27 (0) | 17.48 (0) | 40.23 (14.76) | 57.03 (18.79) | 67.96 (21.47) | 68.15 (19.74)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 72.71 (0) | 20.70 (0) | 51.03 (22.43) | 84.88 (7.67) | 106.0 (44.36) | 137.0 (15.99)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 71.57 (0) | 24.35 (0) | 54.79 (49.63) | 85.71 (16.02) | 103.5 (35.21) | 131.1 (13.87)

12. Secondary Outcome: Plasma Concentration of Glycine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 217.2 (0) | 282.2 (68.99) | 164.4 (0.97) | 188.9 (20.63) | 153.2 (23.80) | 183.2 (16.61)
  Period 1 @ 4.5hrs | 304.6 (0) | 316.8 (113.2) | 243.6 (9.33) | 332.3 (37.75) | 254.0 (8.27) | 417.6 (142.8)
  Period 1 @ 7hrs | 307.1 (0) | 388.4 (63.14) | 248.7 (8.33) | 331.70 (32.97) | 234.5 (13.48) | 477.0 (214.5)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 215.9 (0) | 316.3 (0) | 196.7 (33.50) | 210.1 (45.73) | 162.3 (17.64) | 223.8 (73.09)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 252.0 (0) | 372.3 (0) | 272.2 (50.56) | 394.9 (73.01) | 318.1 (94.07) | 473.2 (194.6)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 278.3 (0) | 409.9 (0) | 272.9 (21.39) | 383.2 (77.85) | 315.0 (48.70) | 481.5 (207.0)

13. Secondary Outcome: Plasma Concentration of Histidine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 59.79 (0) | 68.48 (23.33) | 53.21 (3.43) | 64.81 (11.94) | 60.28 (17.90) | 67.55 (6.56)
  Period 1 @ 4.5hrs | 102.0 (0) | 85.49 (35.85) | 92.18 (6.92) | 127.80 (0.95) | 110.7 (11.70) | 189.8 (65.20)
  Period 1 @ 7hrs | 105.1 (0) | 101.5 (27.27) | 102.0 (5.50) | 134.2 (5.65) | 109.5 (0.79) | 257.0 (157.5)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 57.64 (0) | 82.09 (0) | 49.86 (8.74) | 68.17 (14.31) | 64.02 (3.67) | 73.54 (3.86)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 78.64 (0) | 107.6 (0) | 88.02 (1.17) | 147.5 (12.87) | 131.1 (30.02) | 186.4 (57.07)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 92.85 (0) | 122.2 (0) | 96.02 (6.94) | 166.2 (6.55) | 130.3 (15.85) | 217.7 (99.88)

14. Secondary Outcome: Plasma Concentration of Isoleucine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 78.62 (0) | 44.71 (1.33) | 51.67 (9.86) | 62.79 (4.14) | 58.87 (22.53) | 73.22 (0.92)
  Period 1 @ 4.5hrs | 113.6 (0) | 46.11 (2.99) | 106.6 (12.32) | 111.2 (2.28) | 112.1 (8.92) | 192.9 (68.37)
  Period 1 @ 7hrs | 122.3 (0) | 47.07 (0.78) | 141.5 (25.44) | 116.3 (4.68) | 138.3 (8.17) | 247.5 (122.0)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 61.12 (0) | 44.49 (0) | 77.59 (36.35) | 64.74 (15.58) | 53.35 (30.00) | 76.08 (8.34)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 76.59 (0) | 69.09 (0) | 105.8 (47.35) | 142.9 (17.86) | 127.7 (77.87) | 193.5 (38.50)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 77.31 (0) | 89.49 (0) | 108.9 (72.63) | 181.3 (12.57) | 137.3 (99.68) | 228.1 (64.48)

15. Secondary Outcome: Plasma Concentration of Leucine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 105.0 (0) | 88.40 (1.63) | 88.55 (20.92) | 83.72 (8.61) | 90.14 (30.71) | 124.3 (1.61)
  Period 1 @ 4.5hrs | 144.8 (0) | 76.54 (0.83) | 156.9 (27.03) | 137.8 (0.51) | 157.2 (16.09) | 270.9 (88.68)
  Period 1 @ 7hrs | 150.00 (0) | 71.11 (5.83) | 199.3 (42.32) | 134.0 (18.30) | 180.0 (10.33) | 344.6 (173.9)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 85.48 (0) | 77.60 (0) | 105.3 (64.54) | 84.90 (22.05) | 92.46 (12.77) | 131.0 (8.08)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 98.69 (0) | 112.3 (0) | 130.9 (74.81) | 179.5 (30.22) | 173.9 (83.38) | 277.6 (71.59)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 94.28 (0) | 135.4 (0) | 124.4 (93.67) | 218.6 (9.36) | 186.9 (114.5) | 326.3 (101.7)

16. Secondary Outcome: Plasma Concentration of Lysine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 169.4 (0) | 153.5 (23.62) | 137.8 (9.50) | 152.2 (1.90) | 150.8 (49.38) | 205.8 (37.52)
  Period 1 @ 4.5hrs | 213.8 (0) | 167.4 (6.38) | 208.7 (11.18) | 254.1 (18.31) | 246.0 (25.41) | 396.5 (50.69)
  Period 1 @ 7hrs | 212.2 (0) | 183.2 (41.15) | 224.0 (11.58) | 252.1 (25.75) | 235.10 (16.79) | 461.7 (109.8)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 160.6 (0) | 132.0 (0) | 140.6 (17.39) | 154.6 (9.27) | 157.6 (29.60) | 234.4 (3.42)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 189.7 (0) | 172.5 (0) | 203.2 (15.35) | 289.3 (15.13) | 279.6 (95.81) | 429.3 (69.88)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 205.3 (0) | 206.8 (0) | 209.7 (45.73) | 303.8 (49.51) | 278.3 (105.0) | 437.7 (56.65)

17. Secondary Outcome: Plasma Concentration of Methionine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 22.79 (0) | 20.33 (2.29) | 17.88 (1.83) | 21.20 (0.23) | 15.96 (4.54) | 23.39 (0.55)
  Period 1 @ 4.5hrs | 53.19 (0) | 35.06 (3.34) | 56.60 (2.19) | 77.47 (9.77) | 58.39 (5.08) | 132.5 (57.06)
  Period 1 @ 7hrs | 61.44 (0) | 48.44 (3.80) | 69.93 (1.00) | 99.33 (7.30) | 64.98 (12.04) | 218.50 (140.3)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 19.18 (0) | 28.76 (0) | 18.35 (1.83) | 20.07 (0.15) | 15.98 (4.09) | 26.73 (6.80)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 43.63 (0) | 47.99 (0) | 54.89 (1.38) | 86.24 (3.05) | 82.96 (31.71) | 127.9 (52.59)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 53.57 (0) | 62.97 (0) | 69.01 (9.43) | 177.2 (18.41) | 103.8 (45.25) | 186.6 (100.9)

18. Secondary Outcome: Plasma Concentration of Ornithine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 65.99 (0) | 56.25 (6.89) | 48.50 (6.93) | 36.15 (2.64) | 62.47 (1.51) | 72.31 (0.38)
  Period 1 @ 4.5hrs | 76.46 (0) | 53.26 (6.92) | 74.83 (6.75) | 52.15 (2.32) | 94.60 (18.24) | 117.0 (22.25)
  Period 1 @ 7hrs | 73.94 (0) | 60.75 (10.88) | 111.3 (7.29) | 70.69 (2.96) | 111.1 (22.55) | 183.1 (70.92)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 44.10 (0) | 53.40 (0) | 55.20 (0.77) | 45.40 (2.81) | 66.82 (11.00) | 71.57 (14.10)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 47.40 (0) | 63.29 (0) | 68.22 (13.24) | 69.56 (5.56) | 91.27 (0.83) | 104.6 (15.46)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 53.58 (0) | 80.14 (0) | 81.59 (36.61) | 97.83 (16.31) | 113.3 (29.62) | 145.1 (8.72)

19. Secondary Outcome: Plasma Concentration of Phenylalanine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 64.83 (0) | 62.14 (9.96) | 63.96 (1.48) | 77.74 (53.20) | 58.07 (8.79) | 70.80 (2.72)
  Period 1 @ 4.5hrs | 105.8 (0) | 79.75 (0.39) | 117.4 (5.35) | 164.8 (64.84) | 113.5 (3.73) | 205.6 (71.52)
  Period 1 @ 7hrs | 119.6 (0) | 106.2 (22.37) | 147.3 (4.97) | 220.4 (103.1) | 122.6 (13.89) | 303.6 (158.2)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 59.96 (0) | 65.00 (0) | 56.40 (2.80) | 83.63 (49.38) | 56.96 (2.38) | 71.17 (10.26)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 91.84 (0) | 86.46 (0) | 106.5 (1.20) | 182.4 (80.49) | 137.90 (33.42) | 191.7 (56.38)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 107.3 (0) | 99.77 (0) | 128.3 (18.08) | 248.7 (120.2) | 160.5 (47.84) | 253.0 (94.40)

20. Secondary Outcome: Plasma Concentration of Proline
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 231.3 (0) | 131.9 (39.20) | 126.4 (31.64) | 182.8 (49.00) | 177.0 (73.16) | 216.5 (45.65)
  Period 1 @ 4.5hrs | 270.9 (0) | 135.5 (36.88) | 201.6 (40.98) | 285.5 (25.26) | 275.2 (43.89) | 412.0 (57.04)
  Period 1 @ 7hrs | 268.5 (0) | 146.0 (21.91) | 243.8 (54.40) | 297.8 (33.74) | 284.3 (24.20) | 501.8 (151.6)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 161.6 (0) | 212.5 (0) | 135.5 (21.04) | 230.9 (9.20) | 183.2 (76.25) | 256.3 (34.95)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 186.2 (0) | 264.5 (0) | 202.0 (46.23) | 372.2 (13.29) | 315.6 (131.3) | 454.2 (113.5)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 206.5 (0) | 271.4 (0) | 228.2 (97.49) | 399.0 (23.65) | 331.3 (158.1) | 506.5 (150.2)

21. Secondary Outcome: Plasma Concentration of Serine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 112.70 (0) | 92.46 (0.25) | 77.91 (8.55) | 97.72 (6.94) | 76.12 (6.26) | 76.13 (10.25)
  Period 1 @ 4.5hrs | 142.0 (0) | 92.09 (14.88) | 112.0 (3.11) | 144.0 (15.52) | 130.2 (24.73) | 162.6 (37.36)
  Period 1 @ 7hrs | 148.7 (0) | 107.9 (3.32) | 121.9 (7.28) | 139.5 (8.22) | 120.7 (32.39) | 193.1 (79.13)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 110.0 (0) | 114.3 (0) | 88.03 (12.96) | 102.7 (6.77) | 77.26 (9.07) | 100.9 (8.89)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 107.8 (0) | 132.7 (0) | 105.1 (7.08) | 170.6 (14.82) | 123.6 (11.21) | 192.3 (51.81)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 118.0 (0) | 155.4 (0) | 109.6 (25.36) | 165.1 (30.39) | 126.5 (5.98) | 211.2 (75.94)

22. Secondary Outcome: Plasma Concentration of Taurine
Time Frame: Three times during each 7 hour visit
Population: No data available as no data for this outcome measure were collected during the study.
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Plasma Concentration of Threonine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 209.6 (0) | 93.40 (29.19) | 79.93 (35.53) | 119.5 (16.03) | 100.2 (39.51) | 154.2 (24.56)
  Period 1 @ 4.5hrs | 266.7 (0) | 94.60 (37.36) | 129.1 (27.90) | 181.3 (40.39) | 160.1 (26.40) | 290.7 (118.3)
  Period 1 @ 7hrs | 260.7 (0) | 107.5 (24.62) | 161.6 (37.56) | 202.6 (35.70) | 162.5 (16.42) | 362.0 (197.0)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 208.7 (0) | 121.9 (0) | 94.87 (27.61) | 128.8 (22.22) | 111.7 (4.21) | 176.6 (61.58)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 210.6 (0) | 152.3 (0) | 135.2 (31.78) | 222.4 (29.51) | 193.7 (45.62) | 337.9 (146.8)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 223.6 (0) | 183.8 (0) | 148.4 (55.95) | 248.5 (71.49) | 211.4 (75.37) | 363.8 (179.8)

24. Secondary Outcome: Plasma Concentration of Tyrosine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 78.10 (0) | 67.08 (22.47) | 58.22 (3.82) | 60.28 (14.06) | 51.25 (10.35) | 85.15 (14.45)
  Period 1 @ 4.5hrs | 71.64 (0) | 53.42 (16.60) | 63.50 (6.52) | 60.03 (9.87) | 58.22 (7.83) | 86.43 (19.95)
  Period 1 @ 7hrs | 60.88 (0) | 54.88 (25.08) | 62.50 (5.36) | 51.26 (5.37) | 52.90 (5.96) | 80.88 (24.13)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 64.19 (0) | 66.48 (0) | 53.81 (4.30) | 67.60 (4.60) | 55.68 (8.37) | 88.24 (25.57)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 55.47 (0) | 67.91 (0) | 50.02 (3.79) | 73.08 (0.53) | 58.20 (17.76) | 99.76 (32.81)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 54.80 (0) | 78.05 (0) | 44.42 (7.00) | 71.62 (8.59) | 52.24 (20.36) | 105.4 (46.80)

25. Secondary Outcome: Plasma Concentration of Valine
Time Frame: Three times during each 7 hour visit
Population: One subject completed Period 1, but withdrew from the study prior to the start of Period 2.
Measure: Mean (Standard Deviation); unit: micromol/L
Arm/Group | 15% CLINISOL 0.04 g/kg/hr (AB) | 15% CLINISOL 0.04 g/kg/hr (BA) | 15% CLINISOL 0.08 g/kg/hr (AB) | 15% CLINISOL 0.08 g/kg/hr (BA) | 15% CLINISOL 0.13 g/kg/hr (AB) | 15% CLINISOL 0.13 g/kg/hr (BA)
Number analyzed (Participants) | 1 | 2 | 2 | 2 | 2 | 2
micromol/L
  Period 1 @ 3hrs | 187.6 (0) | 165.6 (11.94) | 159.6 (44.44) | 171.7 (9.35) | 179.8 (45.09) | 245.5 (3.68)
  Period 1 @ 4.5hrs | 257.6 (0) | 167.8 (22.42) | 260.2 (50.23) | 282.0 (8.70) | 296.2 (15.89) | 477.7 (125.8)
  Period 1 @ 7hrs | 281.1 (0) | 186.6 (4.18) | 356.2 (63.52) | 332.7 (27.59) | 353.9 (17.09) | 663.9 (260.3)
  Period 2 @ 3hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 3hrs | 177.1 (0) | 136.7 (0) | 177.5 (88.16) | 177.4 (38.16) | 199.1 (7.82) | 264.2 (11.62)
  Period 2 @ 4.5hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 4.5hrs | 208.4 (0) | 188.7 (0) | 247.3 (110.0) | 323.7 (45.42) | 338.1 (84.89) | 480.9 (71.82)
  Period 2 @ 7hrs: number analyzed (Participants) | 1 | 1 | 2 | 2 | 2 | 2
  Period 2 @ 7hrs | 230.1 (0) | 248.4 (0) | 241.1 (226.3) | 433.4 (31.96) | 399.8 (178.2) | 635.1 (159.6)

ADVERSE EVENTS:
Description: AE analysis provided for all subjects who were exposed to study treatment.
Arm/Group | 15% CLINISOL 0.04 g/kg/hr | 15% CLINISOL 0.08 g/kg/hr | 15% CLINISOL 0.13 g/kg/hr
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/3 | 0/4 | 0/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 15% CLINISOL 0.04 g/kg/hr (N=3) | 15% CLINISOL 0.08 g/kg/hr (N=4) | 15% CLINISOL 0.13 g/kg/hr (N=4)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other